CLINICAL TRIAL: NCT03432117
Title: Multicenter Prospective Clinical Trial to Evaluate Efficacy of Respiratory Rehabilitation Personalized Mobile Services for Respiratory Diseases
Brief Title: Evaluate Efficacy of Respiratory Rehabilitation Personalized Mobile Services for Respiratory Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Ministry of Trade, Industry and Energy (Unknown); Lifesemantics Corp. (Industry)
Responsible Party: Principal Investigator, Chang-Min Choi, associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C2016-00568
Record Dates: First submitted 2018-01-22; First posted 2018-02-14 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Respiratory Disease; Lung Cancer; COPD
Keywords: respiratory rehabilitation; personalized mobile services
MeSH Terms: conditions — Respiration Disorders; Lung Neoplasms; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The subjets were randomized(1:1:1) to 3 group(A: Fixed respiratory rehabilitation program group, B: Mixed respiratory rehabilitation program group( Fixed respiratory rehabilitation for 6 weeks, and then responsive respiratory rehabilitation for 6 weeks) and C: Control group(Ordinary rehabilitation service of the site).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fixed respiratory rehabilitation program(A) (Experimental): respiratory rehabilitation program for 12 weeks
  Interventions: Other: Fixed respiratory rehabilitation
- Mixed respiratory rehabilitation program(B) (Experimental): Fixed respiratory rehabilitation for 6 weeks, and then responsive respiratory rehabilitation for 6 weeks
  Interventions: Other: Fixed respiratory rehabilitation; Other: Responsive respiratory rehabilitation
- Control(C) (No Intervention): Ordinary rehabilitation service of the site for 12 weeks

INTERVENTIONS:
Other: Fixed respiratory rehabilitation — There are 6 step-exercise presented in the application and initial target of exercise will be set according to subject condition. After subject completes targeted exercise, next step will be started.
  Arms: Fixed respiratory rehabilitation program(A); Mixed respiratory rehabilitation program(B)
Other: Responsive respiratory rehabilitation — The application provide responsive exercise program by changing type and numbers of exercise according to subject condition and exercise ability (This will be assessed with monitored O2 saturation, symptom of dyspnea and pulse rate during exercise)
  Arms: Mixed respiratory rehabilitation program(B)

SUMMARY:
This trial is multicenter prospective study to evaluate clinical efficacy of respiratory rehabilitation personalized mobile services for respiratory disease.

DETAILED DESCRIPTION:
Patients with Lung Cancer or COPD who need respiratory rehabilitation were enrolled in this trial. The subjets were randomized to 3 group(A: Fixed respiratory rehabilitation program group, B: Mixed respiratory rehabilitation program group(Fixed respiratory rehabilitation for 6 weeks, and then responsive respiratory rehabilitation for 6 weeks) and C: Control group(Ordinary rehabilitation service of the site)).

Patients in Group A&B were provided with mobile application and wearable O2 saturation machine and mobile application monitors physical activity and provides

1. how to do stretching, weight training with The-ra Band
2. daily and weekly target of exercise
3. alarm algorithms depending on patient's respiratory status(purse rate and O2 saturation)

ELIGIBILITY:
Inclusion Criteria:

* Patients with Lung cancer or COPD
* Patients with FEV1<80% or FVC<80% in Pulmonary function test

  * In case of COPD, post-bronchodilator FEV1 or FVC will be used.
  * Exceptionally Lung Cancer patients with operation, FEV1>80% or FVC>80% will be permitted
* The distance walked for 6 minutes in 6-minute walk test ≥ 150 m
* Patients with android phone
* Patients who voluntarily agree to study participation and provide written informed consent form

Exclusion Criteria:

* Patients with diseases which could be cause of death or significant disability for 1 year after study enrollment.
* Patients with diseases that are difficult to walk or improve walking at screening
* Patients with significant diseases which are difficult to include in this study in accordance with the investigator's judgment
* Patients who are illiterate or have communication limitations
* Patients who have a difficulty to complete a questionnaire or are uncooperative due to deterioration of recognition function

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2018-01-06 (Actual)

PRIMARY OUTCOMES:
change from baseline in Modified Medical Research Council dyspnea score | 12 weeks
  The MMRC dyspnea scale is a five-option grading system. The scale measures a person's limitation base on a scale of 0-4 and uses the final value to determine how much disability is caused by shortness of breath.
change from baseline in COPD Assessment Test(CAT) score | 12 weeks
  The CAT is a validated, short and simple subject completed questionnaire which has been developed for use in routine clinical practice to measure the health status of subjects with COPD. Subjects are scored on eight items (cough, phlegm, chest tightness, breathlessness, activity limitation, confidence, sleep and energy) on a scale of 0-5 depending on their impact. The sum of scores for each item gives the subject's impact score ranging from 0 (no impact) to 40 (worst possible impact).
change from baseline in real distance walked for 6 minutes | 12 weeks

SECONDARY OUTCOMES:
change from baseline in Physical activity | 12 weeks
  Physical activity will be assessed with the daily walking distance monitored by the application and wearable device.
subject satisfaction with health status | 12 weeks
  changed from baseline in EQ-5D-5L
subject satisfaction with service | 12 weeks
  Assessment tool: Patient's Global Assessment - Subjects are scored on four items (general, easy-to-follow, helpful in exercise and Physical fitness ) on a scale of 1-5 depending on their satisfaction level. The sum of scores for each item will be used for assessement of the subject's satisfaction in the trial.
change in Healthcare resource utilisation(the number of hospitalization) in COPD(chronic obstructive pulmonary disease) Patients | 12 weeks
  Comparison with the number of hospitalization during the same period last year
change in Healthcare resource utilisation(hospitalization period) in COPD(chronic obstructive pulmonary disease) Patients | 12 weeks
  Comparison with hospitalization period during the same period last year
change in Healthcare resource utilisation(the number of visiting emergency room) in COPD(chronic obstructive pulmonary disease) Patients | 12 weeks
  Comparison with the number of visiting emergency room during the same period last year

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - KyungHee University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Smg-Snu Boramae Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- [Derived] Kwon H, Lee S, Jung EJ, Kim S, Lee JK, Kim DK, Kim TH, Lee SH, Lee MK, Song S, Shin K. An mHealth Management Platform for Patients with Chronic Obstructive Pulmonary Disease (efil breath): Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Aug 24;6(8):e10502. doi: 10.2196/10502. PMID 30143475